CLINICAL TRIAL: NCT03766269
Title: Dose-Titration Study to Evaluate the Opioid-Sparing Effect of Dronabinol When Coadministered With Opioid Analgesics to Chronic Pain Patients
Brief Title: Dronabinol Opioid Sparing Evaluation (DOSE) Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daisy Pharma Opioid Venture, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 140635
Record Dates: First submitted 2018-11-30; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Dronabinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Baseline Opioid (Other): One of Seven existing Baseline Opioid subgroups (Hydrocodone, Oxycodone, Morphine, Hydromorphone, Buprenorphine, Tramadol) coadministered with intervention drug, Dronabinol.
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — Dronabinol coadministered with patient's existing Baseline Opioid.
  Other Names: Marinol

SUMMARY:
This study will be a 12-week, open-label trial that is designed to evaluate the Opioid-Sparing effect of Dronabinol at ranging doses when coadministered with the opioid analgesics that are currently being prescribed to patients for their chronic pain condition. The purpose of this trial will be to assess the effectiveness of Dronabinol when combined with opioid analgesics to relieve pain at lower opioid doses and to evaluate any reduction of opioid-related side effects. Participants will take the study-drug, Dronabinol, along with their regular prescribed opioids and the results will be evaluated and analyzed according to defined endpoints.

DETAILED DESCRIPTION:
Week one of the study is a Baseline Period during which time, baseline data related to opioid dose and frequency, mood, sleep, bowel movements, and pain intensity will be collected. Participants will receive no Dronabinol during week one and will continue to take their stabilized dose of regular prescribed opioids, both baseline and rescue.

Weeks two through four is the Titration Period, during which time study participants will titrate the Dronabinol dose up to a daily dose of 20 mg of Dronabinol per day, according to a prearranged titration table. Participants will continue to take their stabilized dose of regular prescribed opioids, both baseline and rescue. Participants will be encouraged to maintain the 20mg daily total dose of Dronabinol. Participants may also reduce their dose of Dronabinol at any time (if they experience severe adverse effects) to a minimum daily dose of Dronabinol of 10mg per day. Participants who cannot tolerate at least a minimum daily dose of 10mg of Dronabinol per day will be discontinued from the study.

Weeks five through twelve is the Opioid-Sparing Period, during which time participants will be encouraged to maintain the stabilized dose of Dronabinol that they "found" during the Study-Drug Dose Finding Period. Study Participants will continue to take their regular prescribed opioids, but will be encouraged to reduce their opioid dose and/or opioid dose frequency at any time during the remainder of the study should they experience a reduction in pain and/or an improvement in opioid-related side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read, speak, and understand English;
2. Provision of signed and dated informed consent form;
3. Stated willingness to comply with all study procedures and availability for the duration of the study;
4. Male, Female, or Transgender aged > 18;
5. In fair and stable general health as evidenced by medical history and physical examination, and confirmed by prescriber;
6. Participants who have been diagnosed with a pain condition that has not adequately responded to other treatments, in the judgement of the provider;
7. Participants who are currently taking a stabilized dose of opioid analgesics, and who have been taking opioid analgesics for at least 3-months, and who report a score of > 3 on the Brief Pain Inventory 0-10 severity index.;
8. Ability to take medications as prescribed and willingness to adhere to the study-drug regimen;
9. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to enrollment and agreement to use such a method during study participation;
10. Agreement to abstain from the use of cannabis or other cannabinoid compounds, other than the study-drug Dronabinol, throughout study duration;

Exclusion Criteria:

1. Current substance abuse by self-report;
2. Current use of cannabis or other cannabinoid compounds;
3. Significant baseline nausea, vomiting, sedation, or other symptoms reported by physician and or patient that may compromise the collection of study-related data;
4. A history of seizures, head trauma, and or mental illness ;
5. Pregnancy or lactation;
6. Known allergic reactions to components of Dronabinol;
7. Taking any of the following drugs:

Strong CYP2C9 Inhibitor (e.g., amiodarone, fluconazole) Strong CYP3A4 Inhibitor (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, erythromycin) Potent CYP2C9 or CYP3A4 inducers (e.g., rifampicin) Drugs that are highly protein-bound (e.g., warfarin, cyclosporine, amphotericin B)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Scale (0-10) | Daily (Days 1-82)
  To measure the change in pain intensity from baseline using the Opioid Sparing Diary Toolkit. The measurement of the pain intensity will be derived from the Brief Pain Inventory (Short-Form) item #3. "Please rate your pain by marking the box beside the number that best describes your pain at its worst in the last 24 hours." The score is reported as a value between 0 and 10, with 0 indicative of no pain, and 10 indicative of "pain as bad as you can imagine". The score will be considered a continuous level of measurement.
Self-Reported Opioid Use (Opioid Dose) | Daily (Days 1-82)
  To measure the change in opioid dose from baseline using the Opioid Sparing Diary Toolkit
Self-Reported Opioid Use Frequency (Opioid Dose Frequency) | Daily (Days 1-82)
  To measure the change in opioid use frequency from baseline using the Opioid Sparing Diary Toolkit

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To evaluate and measure any changes in pain history, intensity, location, relief, and life interference indicators from baseline
Hospital and Anxiety Depression Scale (HADS) | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To measure the change in depression and generalized anxiety from baseline. The HADS measures levels of anxiety and depression that a patient is experiencing. The HADS is a fourteen item scale. Seven of the items relate to a factor that measures anxiety and seven relate to a factor that measures depression. The seven items for each factor are summed into a total score and range from 0 to 21, with higher scores indicative of greater anxiety/depression. The scores will be analyzed as continuous level variables and one-sided paired-samples t-tests will be used to compare mean scores for anxiety and depression for all subjects between Week 1 (baseline) and Week 12 (EOS).
Side Effect Checklist 29-item | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To evaluate the presence or absence of side effects associated with the intervention
RAND Health Survey 36-item | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To measure the change in overall quality of life from baseline
MOS Sleep Scale | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To measure the change in quality of sleep from baseline. The MOS Sleep Scale Self Report includes 12 items which measure 7 individual continuous-level factors relating to sleep quality: (a) sleep disturbances, (b) snoring, (c) sleep short of breath or headache, (d) sleep adequacy, (e) sleep somnolence, (f) sleep problems index I, and (g) sleep problems index II. Each of the seven factors is scored via a two-step process such that higher resulting scores are indicative of greater sleep problems. All 7 scores are measured at the continuous level.
Treatment Satisfaction Questionnaire for Medication (TSQM) | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To measure the change in satisfaction with medication from baseline
Bowel Function Inventory-Revised (BFI-R) | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To measure the change in Opioid-Induced Constipation from baseline
Current Opioid Misuse Measure (COMM) | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To measure the change in Possible Opioid Misuse from baseline
Numerical Opioid Side Effect (NOSE) Assessment | Study Visits 1-5 (Days 1, 14, 28, 56, 82)
  To measure the change in Opioid Side Effect Severity from baseline
OSD: Mood Scale Self Report (0-10) | Daily (Days 1-82)
  To measure the change in Mood from baseline. The Mood Scale is a 10 item Likert-scaled instrument with each of the 10 items scored from 1 = absolutely miserable to 10 = absolutely happy. The scores for each of the 10 items will be summed into a mood total score. The mood total score can range from 10 to 100, with higher scores indicative of happier states. The mood total score is a continuous level of measurement.
OSD: Sleep Scale Self Report (0-10) | Daily (Days 1-82)
  To measure the change in Quality of Sleep from baseline. The Sleep Scale is a 10 item Likert-scaled instrument with each of the 10 items scored from 1 = worst imaginable to 10 = best . The scores for each of the 10 items will be summed into a sleep total score. The sleep total score can range from 10 to 100, with higher scores indicative of better quality sleep. The sleep total score is a continuous level of measurement.
OSD: Bowel Movement 24-Hour Self Report Survey | Daily (Days 1-82)
  To measure the change in number of Bowel Movements from baseline
FITBIT: Sleep Tracker | Daily (Days 1-82)
  To measure the change in quantity and quality of sleep from baseline
FITBIT: Distance Tracker | Daily (Days 1-82)
  To measure the change in average weekly distance traveled from baseline
FITBIT: Caloric Expenditure Tracker | Daily (Days 1-82)
  To measure the change in average weekly calories expended from baseline
Medical Billing Claims Data for each participant | Study Visits 1 & 5 (Days 1 & 82)
  To evaluate the change in Health Care Expenditures Related To Chronic Pain from baseline (average monthly expenditures before study)

CONTACTS AND LOCATIONS:
Overall Officials: Kendric B Speagle, BA, Principal Investigator — Daisy Research
Locations (1):
- Daisy Research, Inc., Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided